CLINICAL TRIAL: NCT04077528
Title: Research on Severe Asthma
Acronym: RAMSES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18033J; 2018-A03282-53 (Registry Identifier: Numeber IDRCB)
Record Dates: First submitted 2019-07-15; First posted 2019-09-04 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Adult Severe Asthma Patients Treated in France
Keywords: Severe asthma; Adult; Respiratory disease
MeSH Terms: conditions — Asthma; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The French Society for Respiratory diseases (SPLF), through its Asthma and Allergy working group (G2A), wishes to set up a national cohort of severe asthma patients to describe this population and the use of step 4 and 5 treatment. This study also meets the demand for post - registration studies required by the Health Authorities for biotherapies and bronchial thermoplasty.

Other European or international cohorts of asthmatic patients exist and RAMSES could contribute to data sharing initiatives.

DETAILED DESCRIPTION:
Severe asthma is defined by poorly controlled disease despite treatment with high doses of inhaled corticosteroids, in combination with at least a long acting beta agonist, after optimal management for at least 6 months by an asthma specialist. The diagnosis of severe asthma can only be made after a rigorous evaluation of 6 to 12 months, including the review of diagnosis and treatment, by a pulmonologist, to distinguish difficult asthma from severe asthma.

Severe asthma accounts for 3.5% to 5% of all asthma patients, a population estimated at 150 000 patients in France. This disease is responsible for significant health costs related to asthma treatments, comorbidities, hospitalizations and sick days. The management of severe asthma is complex, multidisciplinary and includes drug treatment, but also the management of side effects of treatment, including oral corticosteroid therapy, and comorbidities of asthma.

Until 2018, omalizumab,systemic continuous oral corticosteroid therapy or inclusion in a therapeutic trial were the ony possibilities offered to severe asthmatic patients beyond the usually recommended and optimized management. In 2018, mepolizumab and reslizumab have been marketed in France, then benralizumab in 2019. They will probably be followed by dupilumab and bronchial thermoplasty. New initiatives to change the history of the disease are also proposed such as specific immunotherapy or long-term use of macrolides. Respiratory rehabilitation is also part of the treatments to be evaluated in some groups of patients.

The description of the use of these treatments, as well as the evaluation of their effectiveness and tolerance in real life conditions is essential. Indeed, their use outside clinical trials raises a number of issues such as the optimal duration of treatment, the maintenance of efficacy over extended periods, the risk and the time to relapse when the treatment is stopped, the possibility to switch from one biotherapy to another in case of insufficient clinical response or to associate them which may prove to be an effective strategy in patients eligible for two biotherapies (allergic and eosinophilic patients).

The cost of these treatments is high. The pharmaco-economic evaluation of severe asthma and its management is another important element. For example, no economic evaluation of the use of omalizumab is currently available in France.

Lastly, the organization of a care network dedicated to severe asthma is being launched in France (severe asthma centers ), on the model of European countries, in order to improve the diagnosis and management of these patients and to reduce the burden of comorbidities of asthma and steroids side effects.It is therefore essential to set up a clinical research structure that will make it possible to obtain clinical data on this population of severe asthma patients and to evaluate all medical practices in real life conditions.

ELIGIBILITY:
Inclusion Criteria:

- Patient with severe asthma : Meeting the definition of ATS-ERS: which requires a combination of high dose CSI and B2LDA.

Or receiving level 5 support (initiating treatment or already treated) :

* Long-term oral corticosteroids (> 6 months in the year prior to inclusion)
* And / or monoclonal antibody
* And / or bronchial thermoplasty
* And / or other complex costs corresponding to the level 5 treatments

  * Consultant or hospitalized in one of the centers participating in RAMSES study

Exclusion Criteria:

* Patient does not accept the recording of his data in the cohort
* Patient not benefiting from health insurance coverage
* Patient under curatorship or tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult severe asthma patients treated in France
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving asthma treatment | Previous treatment, collected at baseline
  Severe asthma medication (high dose inhaled corticosteroids / B2LDA, Anti IgE antibody, Anti IL5 antibody, daily oral steroids…); Other asthma medications (long acting anticholinergics, montelukast, theophylline, inhaled corticoids); bronchial thermoplasty.
Dose of severe asthma treatments | At baseline
  Severe asthma medication (high dose inhaled corticosteroids / B2LDA, Anti IgE antibody, Anti IL5 antibody, daily oral steroids…)
Duration of asthma treatments | Previous treatment, collected at baseline
  Severe asthma medication (high dose inhaled corticosteroids / B2LDA, Anti IgE antibody, Anti IL5 antibody, daily oral steroids…); Other asthma medications (long acting anticholinergics, montelukast, theophylline, inhaled corticoids); bronchial thermoplasty.
Other medications | At baseline
  Number of patients receiving antidiabetics, Number of patients receiving antidepressants, Number of patients receiving anti-osteoporotic drugs, Number of patients receiving cardiovascular drugs.
Asthma-related comorbidities | At baseline
  Prevalence of asthma related comorbidities such as chronic rhinosinusitis, nasal polyps, gastroesophageal reflux, obesity, obstructive sleep apnea respiratory infections, …
Non-respiratory comorbidities | At baseline
  Prevalence of non-respiratory comorbidities such as osteoporosis, diabetes , cardiovascular diseases...
Asthma control test (ACT) | 12 previous months, collected at baseline
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 items, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). Asthma is controlled when the total score is >20.
Asthma exacerbations | 12 previous months, collected at baseline
  Number of systemic corticosteroids (SC) courses
Forced Expiratory Volume in 1 second (FEV1) | 12 previous months, collected at baseline
  Mean FEV1, expressed in ml.
Number of patients with at least 1 sick leaves due to asthma | 12 previous months, collected at baseline
  Patient-reported sick leaves.
Number of sick leaves due to asthma | 12 previous months, collected at baseline
  Patient-reported sick leaves.
Number of patients with long term disease status for asthma | At baseline
Intensive care unit hospitalization due to asthma exacerbation | During life, collected at baseline
  At least one intensive care unit hospitalization for asthma

SECONDARY OUTCOMES:
Number of unscheduled healthcare visits or hospitalization | At 6 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of patients with unscheduled healthcare visits or hospitalization | At 6 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of unscheduled healthcare visits or hospitalization | At 12 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of patients with unscheduled healthcare visits or hospitalization | At 12 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of unscheduled healthcare visits or hospitalization | At 24 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of patients with unscheduled healthcare visits or hospitalization | At 24 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of unscheduled healthcare visits or hospitalization | At 36 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of patients with unscheduled healthcare visits or hospitalization | At 36 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of unscheduled healthcare visits or hospitalization | At 60 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Number of patients with unscheduled healthcare visits or hospitalization | At 60 months
  Inpatient hospitalizations due to asthma including intensive care unit, inpatient hospitalization for other reasons, emergency department visits and unscheduled ambulatory visits
Daily dose of corticosteroids | At 6 months
  Inhaled corticosteroids, oral corticosteroids (SC) in long term users
Daily dose of corticosteroids | At 12 months
  Inhaled corticosteroids, oral corticosteroids (SC) in long term users
Daily dose of corticosteroids | At 24 months
  Inhaled corticosteroids, oral corticosteroids (SC) in long term users
Daily dose of corticosteroids | At 36 months
  Inhaled corticosteroids, oral corticosteroids (SC) in long term users
Daily dose of corticosteroids | At 60 months
  Inhaled corticosteroids, oral corticosteroids (SC) in long term users
Number of patients with at least 1 other asthma medication | At 6 months
  Long acting beta 2 agonists, long acting anticholinergics, montelukast, macrolides, Anti IgE monoclonal antibodies, theophylline.
Number of patients with at least 1 other asthma medication | At 12 months
  Long acting beta 2 agonists, long acting anticholinergics, montelukast, macrolides, Anti IgE monoclonal antibodies, theophylline.
Number of patients with at least 1 other asthma medication | At 24 months
  Long acting beta 2 agonists, long acting anticholinergics, montelukast, macrolides, Anti IgE monoclonal antibodies, theophylline.
Number of patients with at least 1 other asthma medication | At 36 months
  Long acting beta 2 agonists, long acting anticholinergics, montelukast, macrolides, Anti IgE monoclonal antibodies, theophylline.
Number of patients with at least 1 other asthma medication | At 60 months
  Long acting beta 2 agonists, long acting anticholinergics, montelukast, macrolides, Anti IgE monoclonal antibodies, theophylline.
Asthma exacerbations | 6 months
  Systemic corticosteroids (SC) use or doubling the usual dose or at least 48 hours in SC long term users
Asthma exacerbations | At 12 months
  Systemic corticosteroids (SC) use or doubling the usual dose or at least 48 hours in SC long term users
Asthma exacerbations | At 24 months
  Systemic corticosteroids (SC) use or doubling the usual dose or at least 48 hours in SC long term users
Asthma exacerbations | At 36 months
  Systemic corticosteroids (SC) use or doubling the usual dose or at least 48 hours in SC long term users
Asthma exacerbations | At 60 months
  Systemic corticosteroids (SC) use or doubling the usual dose or at least 48 hours in SC long term users
Number of patients reporting suboptimal treatment adherence | Through study completion, an average of 5 years
  Patient-reported adherence to asthma treatment. Suboptimal treatment is defined as less treatment received than expected.
Drug survival rate | At 6 month
  Proportion of patients still exposed to treatment
Drug survival rate | At 12 months
  Proportion of patients still exposed to treatment;
Time to drug discontinuation | Reported at 6 month
  Median time between the start of treatment and its definitive cessation
Time to drug discontinuation | Reported at 12 month
  Median time between the start of treatment and its definitive cessation.
Asthma control test (ACT) | At 6 months
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 item, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
Asthma control test (ACT) | At 12 months
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 item, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
Asthma control test (ACT) | At 24 months
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 item, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
Asthma control test (ACT) | At 36 months
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 item, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
Asthma control test (ACT) | At 60 months
  Patient-reported asthma symptoms and control will be collected via the ACT questionnaire; a 5 item, self-administered survey that is designed to help the patient describe their asthma and how it affects their daily activities. ACT questionnaire is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
Number of patients with at least 1 sick leaves due to asthma | At 6 months
  Patient-reported sick leaves.
Number of sick leaves due to asthma | At 6 months
  Patient-reported sick leaves.
Number of patients with at least 1 sick leaves due to asthma | At 12 months
  Patient-reported sick leaves.
Number of sick leaves due to asthma | At 12 months
  Patient-reported sick leaves.
Number of patients with at least 1 sick leaves due to asthma | At 24 months
  Patient-reported sick leaves.
Number of sick leaves due to asthma | At 24 months
  Patient-reported sick leaves.
Number of patients with at least 1 sick leaves due to asthma | At 36 months
  Patient-reported sick leaves.
Number of sick leaves due to asthma | At 36 months
  Patient-reported sick leaves.
Number of patients with at least 1 sick leaves due to asthma | At 60 months
  Patient-reported sick leaves.
Number of sick leaves due to asthma | At 60 months
  Patient-reported sick leaves.
St. George's Respiratory Questionnaire (SGRQ) | At 6 months
  The St. George's Respiratory Questionnaire (SGRQ) is a self-reporting questionnaire validated for evaluating quality of life in asthma. The total score is expressed as a percentage, from 0%, no impairment of life quality, to 100%, maximal impairment.
St. George's Respiratory Questionnaire (SGRQ) | At 12 months
  The St. George's Respiratory Questionnaire (SGRQ) is a self-reporting questionnaire validated for evaluating quality of life in asthma. The total score is expressed as a percentage, from 0%, no impairment of life quality, to 100%, maximal impairment.
St. George's Respiratory Questionnaire (SGRQ) | At 24 months
  The St. George's Respiratory Questionnaire (SGRQ) is a self-reporting questionnaire validated for evaluating quality of life in asthma. The total score is expressed as a percentage, from 0%, no impairment of life quality, to 100%, maximal impairment.
St. George's Respiratory Questionnaire (SGRQ) | At 36 months
  The St. George's Respiratory Questionnaire (SGRQ) is a self-reporting questionnaire validated for evaluating quality of life in asthma. The total score is expressed as a percentage, from 0%, no impairment of life quality, to 100%, maximal impairment.
St. George's Respiratory Questionnaire (SGRQ) | At 60 months
  The St. George's Respiratory Questionnaire (SGRQ) is a self-reporting questionnaire validated for evaluating quality of life in asthma. The total score is expressed as a percentage, from 0%, no impairment of life quality, to 100%, maximal impairment.
Asthma Quality of Life Questionnaire (AQLQ) overall score by Visit | At 6 months
  The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions.
Asthma Quality of Life Questionnaire (AQLQ) overall score by Visit | At 12 months
  The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions.
Asthma Quality of Life Questionnaire (AQLQ) overall score by Visit | At 24 months
  The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions.
Asthma Quality of Life Questionnaire (AQLQ) overall score by Visit | At 36 months
  The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions.
Asthma Quality of Life Questionnaire (AQLQ) overall score by Visit | At 60 months
  The AQLQ is a 32-item disease-specific questionnaire that has been designed to measure the functional impairments that are most troublesome to adults with asthma. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale. The overall AQLQ score is the mean response to all 32 questions.
EuroQual 5-Dimension Health Status Questionnaire (EQ-5D) index score and health state assessment | At 6 months
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". Pain/discomfort dimension asks how much pain or discomfort the person has, and anxiety/depression dimension asks how anxious or depressed the person is. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).
EuroQual 5-Dimension Health Status Questionnaire (EQ-5D) index score and health state assessment | At 12 months
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". Pain/discomfort dimension asks how much pain or discomfort the person has, and anxiety/depression dimension asks how anxious or depressed the person is. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).
EuroQual 5-Dimension Health Status Questionnaire (EQ-5D) index score and health state assessment | At 24 months
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". Pain/discomfort dimension asks how much pain or discomfort the person has, and anxiety/depression dimension asks how anxious or depressed the person is. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).
EuroQual 5-Dimension Health Status Questionnaire (EQ-5D) index score and health state assessment | At 36 months
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". Pain/discomfort dimension asks how much pain or discomfort the person has, and anxiety/depression dimension asks how anxious or depressed the person is. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).
EuroQual 5-Dimension Health Status Questionnaire (EQ-5D) index score and health state assessment | At 60 months
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". Pain/discomfort dimension asks how much pain or discomfort the person has, and anxiety/depression dimension asks how anxious or depressed the person is. The respondents self-rate their level of severity for each dimension using three-level (EQ-5D-3L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).
Hospital Anxiety and Depression scale | At 6 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Hospital Anxiety and Depression scale | At 12 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Hospital Anxiety and Depression scale | At 24 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Hospital Anxiety and Depression scale | At 36 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Hospital Anxiety and Depression scale | At 60 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Long term adverse Events associated with corticosteroid therapy. | 60 months
  Frequency of relevant medical events such as osteoporosis, diabetes, cardiovascular disease.
Asthma-related comorbidities | At 6 months
  Prevalence of comorbidities such as rhinosinusitis, obesity, gastroesophageal reflux, sleep obstructive apnea syndrome, …
Asthma-related comorbidities | At 12 months
  Prevalence of comorbidities such as rhinosinusitis, obesity, gastroesophageal reflux, sleep obstructive apnea syndrome, …
Asthma-related comorbidities | At 24 months
  Prevalence of comorbidities such as rhinosinusitis, obesity, gastroesophageal reflux, sleep obstructive apnea syndrome, …
Asthma-related comorbidities | At 36 months
  Prevalence of comorbidities such as rhinosinusitis, obesity, gastroesophageal reflux, sleep obstructive apnea syndrome, …
Asthma-related comorbidities | At 60 months
  Prevalence of comorbidities such as rhinosinusitis, obesity, gastroesophageal reflux, sleep obstructive apnea syndrome, …
Death and cause of death | At 6 months
Death and cause of death | At 12 months
Death and cause of death | At 24 months
Death and cause of death | At 36 months
Death and cause of death | At 60 months
Post-procedural adverse Events associated with bronchial thermoplasty | Up to 24 hours following the procedure
  Frequency of post-procedure medical events such as hemoptysis, respiratory symptoms, asthma, prolonged hospitalization
Post-procedural adverse Events associated with bronchial thermoplasty | From 24 hours to 1 month following the procedure
  Frequency of post-procedure medical events such as hemoptysis, respiratory symptoms, asthma, prolonged hospitalization.
Long term adverse events associated with bronchial thermoplasty | 60 months
  Frequency of long term medical events such as bronchial stenosis.
Events of special interest | From treatment initiation to 3 months following treatment initiation
  Frequency of special interest events including new onset malignancy, severe infection, anaphylaxis.
Events of special interest | From 3 months to 12 months following treatment initiation
  Frequency of special interest events including new onset malignancy, severe infection, anaphylaxis.
Events of special interest | From 3 to 5 years following treatment initiation
  Frequency of special interest events including new onset malignancy, severe infection, anaphylaxis.
Blood eosinophil count | At baseline
Total immunoglobulin E (IgE) | At baseline
Chest computed tomography scan | At baseline
  Dates and description of major findings.
Forced Vital Capacity (FVC) | At baseline
Forced Vital Capacity (FVC) | At 6 months
Forced Vital Capacity (FVC) | At 12 months
Forced Vital Capacity (FVC) | At 24 months
Forced Vital Capacity (FVC) | At 36 months
Forced Vital Capacity (FVC) | At 60 months
Forced Expiratory Volume in 1 second (FEV1) | At 6 months
Forced Expiratory Volume in 1 second (FEV1) | At 12 months
Forced Expiratory Volume in 1 second (FEV1) | At 24 months
Forced Expiratory Volume in 1 second (FEV1) | At 36 months
Forced Expiratory Volume in 1 second (FEV1) | At 60 months
FEV1/FVC ratio | At baseline
FEV1/FVC ratio | At 6 months
FEV1/FVC ratio | At 12 months
FEV1/FVC ratio | At 24 months
FEV1/FVC ratio | At 36 months
FEV1/FVC ratio | At 60 months
RV/TLC ratio | At baseline
RV/TLC ratio | At 6 months
RV/TLC ratio | At 12 months
RV/TLC ratio | At 24 months
RV/TLC ratio | At 36 months
RV/TLC ratio | At 60 months
Fractional exhaled nitric oxide (FENO) | At baseline
Costs of severe asthma management | Through study completion, an average of 5 years
  Total amount of money, expressed in euros, reimbursed by Social Security ( for treatments, medical visits, radiological or laboratory examinations).

CONTACTS AND LOCATIONS:
Overall Officials: Camille TAILLE, MD,PHD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Bichat, Paris, France